CLINICAL TRIAL: NCT02608996
Title: Therapeutic Effects of BNP in Hypertensive Patients
Brief Title: Nesiritide in Hypertension
Acronym: TENSE1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Alessandro Cataliotti, Professor, dr. med., Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-000577-13
Record Dates: First submitted 2015-11-09; First posted 2015-11-20 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Natriuretic Peptide, Brain; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subcutaneous BNP (Active Comparator): Patients will receive gradually increasing doses (10-25 µg/kg) of subcutaneously administered nesiritide (BNP) twice daily for two days, to determine the feasibility, safety and blood pressure lowering effect of BNP so as to identify the optimal dose.
  Interventions: Drug: Nesiritide
- Subcutaneous placebo (Placebo Comparator): Patients will receive subcutaneously administered placebo twice daily for two days for determination of the effect of BNP.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nesiritide — This intervention is designed to determine the optimal dose range of BNP for treatment of patients with uncontrolled hypertension
  Other Names: Natrecor, BNP
  Arms: Subcutaneous BNP
Drug: Placebo — For comparison to elucidate the true effect of nesiritide
  Other Names: Saline solution
  Arms: Subcutaneous placebo

SUMMARY:
Hypertension remains a global burden in cardiovascular disease leading to stroke, myocardial infarction, and heart failure. Its myocardial complications result from increased mechanical load on the heart. Under physiological conditions of increased myocardial load and resulting myocardial stretch, atrial natriuretic peptide (ANP) and B-type natriuretic peptide (BNP) synthesis and secretion occur contributing to maintenance of optimal cardiorenal and blood pressure homeostasis. However, studies indicate that in subjects with cardiovascular diseases the biological structure of these hormones may be altered, thus reducing their favorable protective activities. New studies indicate that early and moderate hypertension is associated with a derangement of the natriuretic peptide system which is characterized by the lack of activation of biologically active ANP and BNP, while severe hypertension is characterized by cardiac release of altered molecular forms of ANP and BNP that have reduced biological properties and/or enhanced degradation.

The broad objective of this proposal is to advance the biology and therapeutics of the NPs with a special focus on the cardiac peptide BNP in human hypertension. Our proposal is based upon the biological properties of BNP (i.e. natriuretic, renin-angiotensin-aldosterone suppressing, vasodilating, anti-fibrotic, anti-hypertrophic and positive lusitropic), its mechanistic role in human hypertension, and thus its potential as an innovative chronic protein therapeutic to enhance the treatment of patients with hypertension. Importantly, BNP is an endocrine hormone normally produced by the human heart, and it has been approved for the treatment of acute heart failure in USA.

ELIGIBILITY:
Inclusion Criteria:

* Office systolic blood pressure (SBP) ≥ 120 mmHg and treatment with at least one anti-hypertensive medication. Unchanged medication regimen the last two weeks prior to inclusion.
* Average day-time SBP > 115 on a 24-h ambulatory BP measurement at screening.

Exclusion Criteria:

* Congestive Heart Failure (any New York Heart Association class)
* Ejection Fraction ≤ 40 %
* Known, not appropriately treated, secondary hypertension
* Myocardial infarction within 3 months of screening
* Unstable angina within 14 days of screening, or any evidence of myocardial ischemia
* Pulmonary hypertension
* Aortic stenosis with maximum jet velocity > 2,5 m/s
* Other valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis or biopsy proven active myocarditis
* Sustained Ventricular Tachycardia or Ventricular Fibrillation within 14 days of screening
* Sustained Atrial Fibrillation
* Second or third degree atrioventricular block without a permanent cardiac pacemaker
* Cerebrovascular event within 3 months of screening, or other evidence of significantly compromised cerebral perfusion
* Proteinuria defined as albumin:creatinine ratio > 100 (equivalent to an excretion of > 1 g/day)
* Nephrotic syndrome
* Body Mass Index > 35
* Total bilirubin of > 25 µmol/L, aspartate aminotransferase or alanine aminotransferase 1.5 times the upper limit of normal range
* Renal insufficiency assessed by estimated glomerular filtration rate (GFR) < 30 ml/min
* Serum sodium of ≤ 135 mmol/L and ≥ 150 mmol/L
* Serum potassium of ≤ 3.5 mmol/L and ≥ 5.5 mmol/L
* Women taking hormonal contraceptives containing estrogens
* Pregnancy
* Patients on prolonged, i.e. more than 30 days, immunosuppressant therapy
* Patients with known, active malignancies
* Patients with orthostatic hypotension
* Participation in a trial with an investigational product within the previous three months
* Any contraindication listed on the Investigator's Brochure of the Investigational Medicinal Product
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure (BP) | 48 hours, from day 1 to day 2. Specifically, it will be assessed before first injection(baseline data) up to 12 hours post last injection.
  Office blood pressure and ambulatory blood pressure monitoring (ABPM) recordings will be used for the analysis

SECONDARY OUTCOMES:
Renal function as assessed by estimated glomerular filtration rate (eGFR) | 48 hours, from day 1 to day 2. Specifically, it will be assessed before first injection (baseline data) up to 12 hours post last injection.
  Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine-cystatin C equation will be used to calculate estimated glomerular filtration rate (eGFR).
Hormonal changes assessed by aldosterone, atrial natriuretic peptide (ANP), N Terminal-ANP, BNP, N Terminal-proBNP, C-type natriuretic peptide and cyclic guanosyl monophosphate. | 48 hours, from day 1 to day 2. Specifically, it will be assessed before first injection (baseline data) up to 12 hours post last injection.
  Will be measured in plasma, and all but aldosterone in urine Collections.
Number of participants with treatment-related adverse events defined as all untoward and unintended responses to the treatment related to any dose administered. | 48 hours, from day 1 to day 2. Specifically, it will be assessed after first injection, up to 12 hours post last injection. A second determination will be done within 3 weeks after last injection (21 days assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Cataliotti, MD, PhD, Principal Investigator — Oslo University Hospital and University of Oslo
Locations (3):
- Norway (3):
  - Oslo University Hopital, Rikshospitalet, Oslo
  - Oslo University Hospital, Ullevål Hospital, Oslo
  - Akershus University Hospital, Strømmen